CLINICAL TRIAL: NCT05050773
Title: A Real-world Study of Clinical Characteristics, Treatment Patterns and Effectiveness in Chinese Patients With Angina Pectoris
Brief Title: Registry Study of Medical Therapy in Patients With Angina Pectoris(GREAT)
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Life oasis public service center (Unknown)
Responsible Party: Principal Investigator, Yong Zeng, Professor and Director, First Ward of Coronary Heart Disease Center, Beijing Anzhen Hospital
Other Study IDs: MEDSCI20210407
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Angina Pectoris; Real World Study
Keywords: Angina Pectoris; Real World Study; Nicorandil
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nicorandil group: Patients who are prescribed with Nicorandil with or without other concomitant medication
- Non-Nicorandil group: Patients who are prescribed with antianginal drugs except Nicorandil

SUMMARY:
The study will be a multi-center, prospective, cohort study based on registration of Chinese angina pectoris patients. After signing the informed consent, all patients will be screened as per the inclusion and exclusion criteria. Estimated 1500 eligible patients will be enrolled. Two natural cohort will be formed according to whether Nicorandil will be prescribed to patients or not. The baseline information of patients will be recorded and patients will be followed up to observe the effectiveness of different anti-angina regimens. Follow-up visits will be conducted at Month 3, 6, 9, 12 after enrollment. The visits at Months 3, 6 and 9 will be conducted in the form of electronic patient reported outcomes (ePRO) + telephone follow-up, and the visit at Month 12 will be conducted on site. Patients are required to fill in the patient diary records (weekly) during the course of the study.

This study is designed to establish a cohort of Chinese angina pectoris patients and compare the effectiveness of different anti-angina regimens in patients with angina pectoris.

DETAILED DESCRIPTION:
After having signed informed consent (Day 0), the patients will be screened for enrollment. About 1500 eligible patients will be enrolled in this study. The basic information of eligible patients including demographic characteristics, history of present illness, past history, Rose questionnaire, vital sign, medication information, SAQ and other optional examination data will be collected at Day 0. At Day 0, the patients will join the study Wechat Mini Program developed for online follow up and patient education by scan the QR code provided by investigators. After enrollment, the following information will be collected by ePRO with WeChat Mini Program or telephone follow up of month 3, 6 and 9: vital sign, medication information, SAQ, AE. The follow up of month 12 will be conducted on site which will collect SAQ, AE and other optional examination data.

ELIGIBILITY:
Inclusion Criteria:

-

1. Patients with angina pectoris who have evidence of coronary angiography or coronary computed tomography angiography (CTA) performed within 1 year and meet any of the following requirements:

1. Imaging examination shows ≥ 50% stenosis and with typical or atypical angina symptoms;
2. Imaging examination shows < 50% stenosis; with typical or similar angina symptoms, and the treadmill exercise test or stress echocardiography or radionuclide stress test results are positive;
3. Post-PCI stenosis of left vessels is ≥ 50%; 2. Currently taking or judged by the physicians as suitable to taking at least one oral antianginal drug (e.g., beta-blockers, nitrates, calcium antagonists and potassium channel openers); 3. Have basic reading and writing abilities, and can correctly fill in the Seattle Angina Questionnaire(SAQ) after being trained by the investigator; 4. Able to use smart phones; 5. Voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Have been diagnosed with malignant tumors that seriously threaten survival and have expected survival time of less than 1 year;
2. Have participated in other clinical studies within the past 1 month;
3. With poor compliance or with other conditions unsuitable for this study as assessed by physicians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: angina pectoris patients
Sampling Method: Probability Sample
Enrollment: 1556 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
SAQ-SS change at Month 12 | at Month 12
  Change in Seattle Angina Questionnaire (SAQ) summary score at Month 12 from baseline

SECONDARY OUTCOMES:
SAQ-SS change at Month 3, 6 and 9 | at Month 3, 6 and 9
  Changes in Seattle Angina Questionnaire (SAQ) summary score at Months 3, 6, and 9 from baseline
Vascular stenosis degree change at Month 12 | at Month 12
  Changes in retest results of vascular stenosis imaging at Month 12 from baseline
Medication compliance | 12 Month
  Medication compliance evaluated by proportion of days covered (PDC)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zeng, MD, Principal Investigator — Anzhen hospital, Capital medical university; Xiliang Zhao, MD, Study Director — Anzhen hospital, Capital medical university
Locations (10):
- China (10):
  - Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Changping District Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Beijing Huaxin Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Miyun District Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Ruyang People's Hospital, Luoyang, Henan
  - Huai'an Hospital of Traditional Chinese Medicine, Huai'an, Jiangsu
  - Dezhou People's Hospital, Dezhou, Shandong

REFERENCES:
- [Derived] Zhao X, Cheng G, Sun L, Liu Y, Du X, Xu S, Wu L, Wei Y, Liu W, Miao L, Zhang Q, Ma C, Zeng Y. Nicorandil Use and Health Status Outcomes in Patients with Angina Pectoris: A Prospective, Multicenter, Cohort Study (GREAT). Drug Des Devel Ther. 2025 Sep 15;19:8295-8308. doi: 10.2147/DDDT.S506108. eCollection 2025. PMID 40980423
- [Derived] Zhao X, Tong Z, Sun L, Zhang Q, Du X, Xu S, Shen C, Wei Y, Liu W, Miao L, Zeng Y. Clinical Characteristics, Treatment Patterns, and Effectiveness in Chinese Patients with Angina Pectoris Using Electronic Patient-Reported Outcomes: Protocol for a Multicenter, Prospective, Cohort Study (GREAT). Adv Ther. 2023 Apr;40(4):1899-1912. doi: 10.1007/s12325-023-02425-0. Epub 2023 Feb 4. PMID 36737594